CLINICAL TRIAL: NCT02432716
Title: A Double-Blind, Placebo-Controlled Pilot Investigation of the Safety of Intranasal Glulisine in Down Syndrome
Brief Title: Investigation of the Safety of Intranasal Glulisine in Down Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HealthPartnersRF
Record Dates: First submitted 2015-04-08; First posted 2015-05-04 (Estimated); Results first posted 2019-12-06 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2018-06

CONDITIONS: Down Syndrome
MeSH Terms: conditions — Down Syndrome | interventions — insulin glulisine; Insulin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Insulin (glulisine), then Placebo (Experimental): Participants first receive one dose of Glulisine 20 IU/IN (.1ml/10 units intranasal in each nostril). After a washout period of 2 weeks, they then received one dose of placebo, Sterile Normal Saline 20 IU/IN (.1ml intransal in each nostril).
  Interventions: Drug: Insulin glulisine; Drug: Saline
- Placebo, then Insulin (glulisine) (Experimental): Participants first receive one dose of placebo, Sterile Normal Saline 20 IU/IN (.1ml intransal in each nostril). After a washout period of 2 weeks, they then received one dose of Glulisine 20 IU/IN (.1ml/10 units intranasal in each nostril).
  Interventions: Drug: Insulin glulisine; Drug: Saline

INTERVENTIONS:
Drug: Insulin glulisine — Insulin (glulisine) Glulisine 20 IU/IN (.1ml/10 units intranasal in each nostril), once per study
  Other Names: insulin, glulisine, Apidra
Drug: Saline — Placebo Comparator: Placebo Sterile Normal Saline 20 IU/IN (.1ml intransal in each nostril), once per study
  Other Names: Placebo

SUMMARY:
This study is a single center, randomized, double-blind, placebo-controlled, cross-over pilot study designed to assess the safety of intranasally (IN) delivered glulisine versus placebo in patients with DS. Subjects will be randomized into this cross-over study and within subject comparisons conducted between single treatment of intranasal insulin glulisine and single treatment of intranasal placebo. All subjects will also receive a single treatment of placebo prior to randomization to ensure adherence to study procedures.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 35-80 years with a Down syndrome diagnosis that is confirmed by karyotype.
* Vital signs must be within normal limits for their age. (Medically treated hypertension will be allowed).
* Must have an electrocardiogram free of clinically significant findings.
* Must have an authorized representative to provide written informed consent.
* Level of speech and comprehension of verbal commands are sufficient to understand and to answer simple requests.
* Must have a reliable caregiver or family member who agrees to accompany the subject to all visits, provide information about the subject as required by this protocol.
* Must be independent for activities of daily living.
* Must tolerate the initial IN treatment of placebo and adhere to study procedures.

Exclusion Criteria:

* Any current psychiatric or neurologic diagnosis other than Down syndrome or Down syndrome with dementia that is judged to impact cognition.
* Subjects who currently meet or have within the past five years met DSM-IV (Diagnostic and Statistical Manual) criteria for drug or alcohol abuse or dependence.
* Subjects residing in a skilled nursing facility or subjects who are anticipated to enter a nursing home within the next 6 months. (Subjects may reside in group homes, assisted living, or other residential settings where they do not require 24 hour skilled nursing.)
* Subjects receiving any experimental drug for Down syndrome within the past 30 days of screening visit.
* Subjects with significant allergies to or other significant intolerance insulin.
* Presence of active seizure disorder.
* Presence of significant aggression or agitation that may impact participation with testing and IN administration. All subjects must have NPI-C aggression and agitation subscore ≤ 4 (severity ≤ 2; frequency ≤ 2).
* Significant cerebrovascular disease with Modified Hachinski Score>4.
* Subjects who may not be able to comply with the protocol or perform the outcomes measures due to significant hearing or visual impairment or other issues judged relevant by the investigators.
* Subject has been diagnosed with any form of diabetes mellitus, actively takes insulin, or has HbA1c > 6.1% at screening.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-04; Primary Completion 2018-10-18 (Actual); Study Completion 2018-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Rosenbloom, MD, Principal Investigator — HealthPartners Institute
Locations (1):
- HealthPartners Neuroscience Center, Saint Paul, Minnesota, United States

REFERENCES:
- [Derived] Rosenbloom M, Barclay T, Johnsen J, Erickson L, Svitak A, Pyle M, Frey W, Hanson LR. Double-Blind Placebo-Controlled Pilot Investigation of the Safety of a Single Dose of Rapid-Acting Intranasal Insulin in Down Syndrome. Drugs R D. 2020 Mar;20(1):11-15. doi: 10.1007/s40268-020-00296-2. PMID 32077057

RESULTS

PARTICIPANT FLOW:
Groups:
- Insulin (Glulisine), Then Placebo: Participants first receive one dose of Glulisine 20 IU/IN (.1ml/10 units intranasal in each nostril). After a washout period of 2 weeks, they then receive one dose of placebo, Sterile Normal Saline 20 IU/IN (.1ml intranasal in each nostril).
- Placebo, Then Insulin (Glulisine): Participants first receive one dose of placebo, Sterile Normal Saline 20 IU/IN (.1ml intransal in each nostril). After a washout period of 2 weeks, they then receive one dose of Glulisine 20 IU/IN (.1ml/10 units intranasal in each nostril).
Period: Overall Study
Arm/Group | Insulin (Glulisine), Then Placebo | Placebo, Then Insulin (Glulisine)
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants first receive either one dose of Glulisine 20 IU/IN (.1ml/10 units intranasal in each nostril) or placebo, Sterile Normal Saline 20 IU/IN (.1ml intranasal in each nostril). After a washout period of 2 weeks, they then receive the opposite.
  Insulin glulisine: Insulin (glulisine) Glulisine 20 IU/IN (.1ml/10 units intranasal in each nostril), once per study
  Saline: Placebo Comparator: Placebo Sterile Normal Saline 20 IU/IN (.1ml intransal in each nostril), once per study
Arm/Group | All Study Participants
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.7 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12
A1C [Mean (Standard Deviation); unit: mmol/mol] | 5.4 (0.1)

OUTCOME MEASURES:

1. Primary Outcome: Safety Measured by Adverse Events
Description: Number of adverse and/or serious events
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin (Glulisine), Then Placebo | Placebo, Then Insulin (Glulisine)
Number analyzed (Participants) | 6 | 6
Participants | 0 | 0

2. Secondary Outcome: Cognitive Change Measured by Fuld Object-Memory Evaluation (FOME)
Description: During the examination, a patient is presented with ten common objects they are asked to identify by touch. The test uses distraction to test recall. For all, a higher score indicates a better outcome.
  * Learning curve is the number of objects the difference in the number of items they are able to correctly identify from the greater of trials 4 or 5 compared to trial 1. Range: 0-10
  * Total immediate recall is the number of objects recalled over all of the trials. Range: 0-50
  * Total delayed recall is the number of objects recalled after 5 minutes. Range: 0-10
  * Recognition memory is the number of items correct from a multiple choice list of three when unable to correctly identify items from delayed recall. Range: 0-10
  * Retention estimate is the number of items recalled after 5 minutes or being reminded with multiple choice. Range: 0-10
Time Frame: 20 minutes
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Post- Placebo: Participants first receive one dose of placebo, Sterile Normal Saline 20 IU/IN (.1ml intransal in each nostril). After receiving intranasal dose, participants completed the Fuld Object-Memory Evaluation.
  Saline: Placebo Comparator: Placebo Sterile Normal Saline 20 IU/IN (.1ml intransal in each nostril), once per study
- Post-Insulin (Glulisine): Participants first receive one dose of Glulisine 20 IU/IN (.1ml/10 units intranasal in each nostril). After receiving intranasal dose, participants completed the Fuld Object-Memory Evaluation.
  Insulin glulisine: Insulin (glulisine) Glulisine 20 IU/IN (.1ml/10 units intranasal in each nostril), once per study
Arm/Group | Post- Placebo | Post-Insulin (Glulisine)
Number analyzed (Participants) | 12 | 12
score on a scale
  Learning Curve | 2.3 (.5) | 2.0 (.6)
  Total Immediate Recall | 33.8 (3.5) | 36.8 (3.3)
  Total Delayed Recall | 6.1 (.6) | 6.4 (.8)
  Recognition Memory | 2.3 (.3) | 1.9 (.5)
  Retention Estimate | 8.3 (.4) | 8.3 (.6)

3. Secondary Outcome: Memory Retention Measured by Fuld Object-Memory Evaluation (FOME)
Description: Memory retention is the percentage of items correctly identify during the delayed recall trial compared storage trial 5. Range: 0-100 percent. A higher percentage indicates a better outcome.
Time Frame: 20 minutes
Measure: Mean (Standard Error); unit: percentage of items correctly identified
Arm/Group | Post- Placebo | Post-Insulin (Glulisine)
Number analyzed (Participants) | 12 | 12
percentage of items correctly identified | 72.3 (5.3) | 68.7 (6.5)

4. Secondary Outcome: Cognitive Change Measured by Rivermead Behavioral Memory Test (RBMT-C)
Description: The RBMT-C provides an objective measure of everyday memory problems reported and observed in subjects with memory difficulties. The test is standardized for use with children ranging in age from 5 to 10 years. Here, we used it for evaluation of Down Syndrome subjects. The story recall subtests involves immediate free recall, cued recall, and delayed recall of short story material which is presented orally to subjects by the examiner. The RBMT-C is appealing for use in this population because the task is engaging, simple, and has been shown in other studies to be an effective measure of memory functions. For all, a higher score means a better outcome.
  * Immediate Recall is the number of story elements recalled right after the story is complete. Range: 0-31
  * Delayed Recall is the number of story elements recalled after a delay. Range: 0-31
Time Frame: 20 minutes
Population: Rivermead Memory Retention is missing for one subject at post-saline time.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Post- Placebo | Post-Insulin (Glulisine)
Number analyzed (Participants) | 12 | 12
score on a scale
  Immediate Recall | 6.6 (1.4) | 5.4 (1.2)
  Delayed Recall | 6.6 (1.5) | 7.2 (1.4)

5. Secondary Outcome: Memory Retention Measured by Rivermead Behavioral Memory Test (RBMT-C).
Description: The RBMT-C provides an objective measure of everyday memory problems reported and observed in subjects with memory difficulties. The test is standardized for use with children ranging in age from 5 to 10 years. Here, we used it for evaluation of Down Syndrome subjects. The story recall subtests involves immediate free recall, cued recall, and delayed recall of short story material which is presented orally to subjects by the examiner. The RBMT-C is appealing for use in this population because the task is engaging, simple, and has been shown in other studies to be an effective measure of memory functions. Memory retention is the percentage of story elements recalled after a delay compared to right after the story is complete. Range: 0-100. A higher score means a better outcome.
Time Frame: 20 minutes
Measure: Mean (Standard Error); unit: percentage of story elements recalled
Arm/Group | Post- Placebo | Post-Insulin (Glulisine)
Number analyzed (Participants) | 12 | 12
percentage of story elements recalled | 9.7 (1.3) | 16.9 (3.8)

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Post-Placebo: Participants first receive one dose of placebo, Sterile Normal Saline 20 IU/IN (.1ml intransal in each nostril). After receiving intranasal dose, participants completed the Fuld Object-Memory Evaluation.
  Saline: Placebo Comparator: Placebo Sterile Normal Saline 20 IU/IN (.1ml intransal in each nostril), once per study
Arm/Group | Post-Placebo | Post-Insulin (Glulisine)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-08-25): https://cdn.clinicaltrials.gov/large-docs/16/NCT02432716/Prot_SAP_000.pdf